CLINICAL TRIAL: NCT01512589
Title: Phase IIB Randomized Trial of Proton Beam Therapy Versus Intensity-Modulated Radiation Therapy for the Treatment of Esophageal Cancer
Brief Title: Proton Beam Therapy (PBT) Versus Intensity-Modulated Radiation Therapy (IMRT) Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1036; NCI-2012-00078 (Registry Identifier: NCI-CTRP-Clinical Trial Reporting Registry); 5U19CA021239 (NIH)
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Cancer
Keywords: Proton Beam Therapy; PBT; Intensity-Modulated Radiation Therapy; IMRT; Esophageal cancer; Adenocarcinoma; Squamous cell carcinoma; Cervical esophagus; Thoracic esophagus; Gastroesophageal junction; Cardia of stomach; Questionnaires; Surveys; Symptom scores; Quality of life; QOL
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Proton Therapy; Radiotherapy; Radiotherapy, Intensity-Modulated; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton Beam Therapy (PBT) (Experimental): Radiation therapy 1 time each day, 5 days a week (Monday through Friday) for up to 28 treatments. 1.8 Gy (or at RBE ("Relative Biologic Equivalence" for PBT)) to be delivered to the periphery of the planning target volume (PTV).
  Interventions: Radiation: Proton Beam Therapy (PBT); Behavioral: Questionnaires
- Intensity Modulated Radiation Therapy (IMRT) (Active Comparator): Radiation therapy 1 time each day, 5 days a week (Monday through Friday) for up to 28 treatments. 1.8 Gy to be delivered to the periphery of the planning target volume (PTV).
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT); Behavioral: Questionnaires

INTERVENTIONS:
Radiation: Proton Beam Therapy (PBT) — 1.8 Gy (Relative Biologic Equivalence ((RBE)) to be delivered to the periphery of the planning target volume (PTV) 1 time each day, 5 days a week (Monday through Friday) for up to 28 treatments.
  Other Names: Radiation Therapy; XRT
  Arms: Proton Beam Therapy (PBT)
Radiation: Intensity Modulated Radiation Therapy (IMRT) — 1.8 Gy to be delivered to the periphery of the planning target volume (PTV) 1 time each day, 5 days a week (Monday through Friday) for up to 28 treatments.
  Other Names: Radiation Therapy; XRT
  Arms: Intensity Modulated Radiation Therapy (IMRT)
Behavioral: Questionnaires — Symptom and Quality of Life questionnaires completed at baseline, every week during radiation therapy, during break after radiation therapy, and during follow up phase.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn how safe and effective proton-beam therapy (PBT) may be in comparison to intensity modulated radiation therapy (IMRT) in combination with chemotherapy in patients with esophageal cancer.

PBT and IMRT are both forms of radiation therapy that are designed to treat a specific area of the body while affecting as little of the surrounding normal tissue as possible. PBT is a newer technology that is designed to further reduce the amount of radiation that affects the surrounding normal tissue. However, this is still being studied.

DETAILED DESCRIPTION:
Study Treatment:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups:

* If you are in Group 1, you will receive IMRT.
* If you are in Group 2, you will receive PBT.

You will receive radiation therapy 1 time each day, 5 days a week (Monday through Friday) for up to 28 treatments.

Your doctor may think it is in your best interest to also receive chemotherapy while you are receiving radiation therapy. If this occurs, you will sign a separate consent form for these drugs with a full description of how they are given and the risks they may cause.

Study Visits:

Before you begin receiving radiation therapy, you will have a baseline visit. The following tests and procedures will be performed:

* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* Your performance status will be recorded.
* You will have a PET/CT or CT scan to check the status of the disease.
* You will have lung function tests
* You will complete the symptom and quality of life questionnaires.
* Your esophagus will be examined using an endoscope. If the doctor thinks it is needed, you will have a biopsy to check the status of the disease.

You will then have a study visit every week while you are receiving radiation therapy. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status, weight, and vital signs will be recorded.
* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* You will complete the symptom and quality of life questionnaires.

Length of Study:

You will receive radiation therapy for up to 28 treatments (about 5½ weeks). You will no longer be able to receive radiation therapy if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the follow-up visits.

Follow-Up:

After you stop receiving radiation therapy, there will be a 4-6 week break. During this time, you will contacted 2 times each week to complete the symptom and quality of life questionnaires. You will receive a call from an automated calling service or from the study staff at a scheduled time of your choosing. You will continue to be followed routinely during treatment and for follow-up visits and tests.

About 4-6 weeks after you stop receiving radiation therapy, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status, weight, and vital signs will be recorded.
* You will have a PET/CT scan to check the status of the disease.
* You will have lung function tests.
* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* You will complete the symptom and quality of life questionnaires.
* Your esophagus will be examined using an endoscope. If the doctor thinks it is needed, you will have a biopsy to check the status of the disease.

If your doctor thinks it is in your best interest after you have completed radiation therapy, you will have surgery to remove the tumor. You will sign a separate consent form that describes the procedure and its risks. As part of this study, the study doctor will check you for side effects and discomfort after the surgery.

Every 3-4 months for 2 years, and then every 4-6 months for the next 3 years, you will have follow-up visits. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status, weight, and vital signs will be recorded.
* You will have either a CT or a PET/CT scan to check the status of the disease.
* You will complete the symptom and quality of life questionnaires. (If the disease gets worse, these questionnaires will no longer be completed.)

Additionally, the following tests and procedures will be performed at follow-up visits only when the doctor thinks they are needed:

* Blood (about 1-2 tablespoons) may be drawn for routine tests.
* You may have lung function tests.
* Your esophagus will be examined using an endoscope. If the doctor thinks it is needed, you will have a biopsy to check the status of the disease.

You may be contacted by the study staff to ask about your health, even if you choose not to return to MD Anderson for follow-up visits after completing treatment for esophageal cancer.

This is an investigational study. IMRT and PBT are delivered using FDA-approved and commercially available methods. It is investigational to compare IMRT to PBT.

Up to 180 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18
2. Histologically documented adenocarcinoma or squamous cell carcinoma of the cervical or thoracic esophagus or gastroesophageal junction or cardia of stomach.
3. Potentially resectable or unresectable esophageal cancer patients
4. Induction chemotherapy prior to concurrent chemoradiation allowed
5. Prior Endoscopic Mucosal Resection (EMR) with a diagnosis of stage II-III esophageal cancer is eligible
6. Performance status of Karnofsky Performance Scale (KPS) >/= 60 or Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2.
7. Prior thoracic radiation allowable only if there is minimal to no overlap with the treatment area estimated at the time of consultation.
8. Negative pregnancy test (serum or urine) for women of child bearing potential. All protocol participants must agree to adequate contraception.
9. Complete blood count (CBC) and complete metabolic panel (chemo-14: Glucose, Calcium, Albumin, Total Protein, Sodium, Potassium, Carbon Dioxide (CO2), Chloride, Blood Urea Nitrogen (BUN), Creatinine, Alkaline Phosphatase, Alanine Aminotransferase (ALT) Serum Glutamic Pyruvic Transaminase (SGPT), Aspartate Aminotransferase (AST) Serum Glutamic-oxaloacetic Transaminase (SGOT), and Bilirubin) to assess adequate hematologic, renal and hepatic functioning will be obtained. The values are as follows: Adequate hematologic (White Blood Count (WBC) >2,500/uL, platelets > 75,000/uL), renal (Serum creatinine </= 1.5X Upper Limit of Normal (ULN) or creatinine clearance > 50 mL/min), and liver function (bilirubin </=1.5 fold the upper limit of normal and liver enzymes < 3 fold the upper limit of normal)
10. Able to communicate in the English language.
11. Any patient deemed eligible for chemoradiation for esophageal cancer treatment.

Exclusion Criteria:

1. Patients with active second malignancy are allowed as long as it is determined by the treating physician that the treatment of esophageal cancer is of higher priority through proper evaluation. However patients with active stage 4, metastatic cancers, receiving other systemic therapies at the time of the esophageal cancer diagnosis, will not be eligible.
2. Pregnant or breast-feeding females
3. Clinically significant uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal or hematologic disease but not limited to: a) active uncontrolled infection; b) Symptomatic congestive heart failure, unstable angina, or cardiac dysrrhythmia not controlled by pacer device; c) no myocardial infarction within 3 months of registration
4. Radiation treatment alone without concurrent chemotherapy or chemotherapy use alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 weeks after radiation therapy
  Defined from the time of enrollment to the date of death or any recurrence. The progression-free survival (PFS) time distribution will be estimated in each treatment arm using the Kaplan-Meier method.
Total Toxicity Burden (TTB) | 12 months
  TTB defined from the time of randomization to 12 months after randomization. Total toxicity burden (TTB) is computed as a composite score from serious adverse events (SAEs) and, among patients who undergo surgery, postoperative complications (POCs).

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Lin, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lin SH, Hobbs BP, Verma V, Tidwell RS, Smith GL, Lei X, Corsini EM, Mok I, Wei X, Yao L, Wang X, Komaki RU, Chang JY, Chun SG, Jeter MD, Swisher SG, Ajani JA, Blum-Murphy M, Vaporciyan AA, Mehran RJ, Koong AC, Gandhi SJ, Hofstetter WL, Hong TS, Delaney TF, Liao Z, Mohan R. Randomized Phase IIB Trial of Proton Beam Therapy Versus Intensity-Modulated Radiation Therapy for Locally Advanced Esophageal Cancer. J Clin Oncol. 2020 May 10;38(14):1569-1579. doi: 10.1200/JCO.19.02503. Epub 2020 Mar 11. PMID 32160096
- See also: M D Anderson Cancer Center — http://www.mdanderson.org